CLINICAL TRIAL: NCT03304717
Title: Reverse Transcriptase Inhibitors in Aicardi Goutières Syndrome
Acronym: RTI in AGS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Results from other clinical trials on AGS established baricitinib as standard of care treatment. Thanks to the knowledge gained in the clinical treatment of AGS, a clinical trial around the effects of RTI in AGS is no longer relevant at this time.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Human Genome Research Institute (NHGRI) (NIH); Gilead Sciences (Industry); Emerson Resources (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-013715; U01HD082806-03 (NIH)
Record Dates: First submitted 2017-08-04; First posted 2017-10-09 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Aicardi Goutières Syndrome
Keywords: Leukodystrophy; Antiretroviral Drugs
MeSH Terms: interventions — Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TDF/FTC then Placebo (Experimental): This is a double-blind, placebo-controlled, 2 arm, cross-over trial involving 34 children with clinical findings and molecular confirmation of Aicardi Goutieres Syndrome, who also have an abnormal interferon signature. For arm 1, half of the patients will receive TDF/FTC (a combination of Tenofovir [TDF] and Emtricitabine [FTC]) for the first 6 months of the study. There will be a one month washout period before starting on placebo for 6 months.
  Interventions: Drug: Tenofovir (TDF) and Emtricitabine (FTC); Other: Placebo
- Placebo then TDF/FTC (Experimental): For arm 2, half of the patients will receive placebo for the first 6 months of the study. There will be a one month washout period before starting on TDF/FTC (a combination of Tenofovir [TDF] and Emtricitabine [FTC]) for 6 months.
  Interventions: Drug: Tenofovir (TDF) and Emtricitabine (FTC); Other: Placebo

INTERVENTIONS:
Drug: Tenofovir (TDF) and Emtricitabine (FTC) — Tenofovir (TDF): a nucleotide reverse transcriptase inhibitor (NtRTI) an acyclic nucleotide analog of adenosine 5'-monophosphate. This is used in children as young as age 2.
  Emtricitabine (FTC): a nucleoside reverse transcriptase inhibitor (NRTI), a synthetic analog of cytidine which binds at the active site of the reverse transcriptase.
  Other Names: Truvada (Tenofovir Disoproxil Fumarate and Emtricitabine); Viread (Brand for tenofovir disoproxil fumarate); Emtriva (Brand for emtricitabine)
Other: Placebo — Placebo for Tenofovir and Placebo for Emtricitabine

SUMMARY:
The overall objectives are to explore the safety and efficacy of Reverse Transcriptase Inhibitors Tenofovir (TDF)/ Emtricitabine (FTC) administered in AGS affected children 2 to 18 years of age.

DETAILED DESCRIPTION:
The investigators propose that a trial to assess the proof of principle that antiretroviral therapy through a drug combination of Tenofovir (TDF) and Emtricitabine (FTC) can decrease endogenous retroelement accumulation, and alter interferon signaling in Aicardi Goutières Syndrome (AGS) patients is reasonable and warranted at this time, based on existing in vitro and animal data. Additionally, this trial will further the investigators understanding of this disorder, measuring for the first time retroelements in human participants, exploring the retroviral burden in cerebrospinal fluid (CSF), the Interferon (IFN) signaling response, as well as evaluating antigen targets of autoimmunity and cytokines. If successful, this approach will clearly demonstrate the need for a larger trial of antiretrovirals in AGS with more clinically relevant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Molecular, neuroimaging, and clinical findings consistent with a diagnosis of AGS, with the exception of Double-stranded RNA-specific adenosine deaminase (ADAR1) and IFIH1, which are not postulated to result in nucleic acid accumulation
* Evidence of interferon activation such as elevation of CSF neopterin/tetrahydrobiopterin measured on the first evaluation.
* Ages 2-18 years (the age of 2 years is used because the drugs are FDA approved in children greater than 2 years)
* Weight of at least 10 kg
* Willingness to undergo serial lumbar punctures and blow draws for evaluation of laboratory based outcome measures
* Willingness to abstain from initiating the use of immune modulating therapies including corticosteroids
* Able to receive medications orally, by nasogastric (NG) tube or by Gastric (G)-tube
* No concomitant illness which would preclude safe participation as judged by the investigator
* Signed informed consent by the subject's legally acceptable representative
* Negative testing for HIV
* Negative testing for Hepatitis B
* Concurrent enrollment in the Myelin Disorders Biorepository Project (MDBP, ClinicalTrials.gov NCT03047369) and willingness to undergo associated procedures

Exclusion Criteria:

* Age < 2 years or >18 years
* Hepatic insufficiency with liver function tests greater than 3-times the upper limit of normal
* Renal insufficiency with creatinine clearance <60
* Significant malabsorption
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at an additional risk by participating in this study
* HIV infection
* Hepatitis B infection
* Mutations in ADAR1 or IFIH1

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in interferon activation as measured by interferon response genes | From Baseline to 13 months
  The investigators propose to measure genes in the IFN stimulatory pathway in AGS patients, as a measure of disease activity and as a possible biomarker of therapeutic activity. Current data suggests that IFN related genes remain elevated in the late teens in AGS affected subjects, making it a more reliable measure of disease activity than IFN alpha. Validation of this preliminary data includes serial measurements in blood across several time points, to assess for variability.

SECONDARY OUTCOMES:
Determination of immune cell composition in CSF | From Baseline to 13 months
  The investigators will pursue immunophenotyping of CSF cells in AGS subjects. Immunophenotyping and target antigens will further understanding of end organ damage in AGS. Additionally, this may provide biomarkers for therapeutic outcome and disease activity.
Determination of immune cell composition in blood | From Baseline to 13 months
  The investigators will pursue immunophenotyping of peripheral blood monocytes in AGS participants. Immunophenotyping and target antigens will further our understanding of end organ damage in AGS. Additionally, this may provide biomarkers for therapeutic outcome and disease activity.
Accumulation of endogenous retroelements as measured in circulating immune cells | From Baseline to 13 months
  Performed by assays from previously collected samples
Accumulation of endogenous retroelements as measured in circulating CSF | From Baseline to 13 months
  Performed by assays from previously collected samples
Change in presence of non-specific and specific autoantibodies in blood | From Baseline to 13 months
  Performed by assays from previously collected samples
Changes in Adverse Events - Safety monitoring laboratory tests | From Baseline to 13 months and as clinically warranted
  Patient monitoring for adverse effects
Changes in total days hospitalized for disease-related illnesses. | Baseline - 13 months
  Assess the effects of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Vanderver, MD, Principal Investigator — Children's Hospital of Philadelphia; William Gahl, MD. PhD, Principal Investigator — National Institute of Health Genome Research Institute